CLINICAL TRIAL: NCT02967393
Title: Feasibility Study to Assess the Safety of Quadrivalent, Live Attenuated Influenza Vaccine (LAIV4) Versus Quadrivalent Inactivated Influenza Vaccine (IIV4) in Children Aged 5-11 Years With Persistent Asthma of Varied Severity (Cell Culture Quadrivalent IIV Used as Surrogate for LAIV4)
Brief Title: Influenza Vaccine Feasibility Study in Children With Persistent Asthma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Duke University (Other); Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, Kathryn Edwards, Sarah H. Sell and Cornelius Vanderbilt Professor of Pediatrics, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IIV4/LAIV4/CDC
Record Dates: First submitted 2016-10-31; First posted 2016-11-18 (Estimated); Results first posted 2018-04-23 (Actual); Last update posted 2018-04-23 (Actual); Status verified 2018-03

CONDITIONS: Asthmatic
MeSH Terms: conditions — Asthma | interventions — Influenza Vaccines; fluarix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IIV4 (Active Comparator): 0.5 mL intramuscular injection
  Interventions: Drug: IIV4
- cc IIV4 (Active Comparator): 0.5 mL intramuscular injection
  Interventions: Drug: ccIIV4

INTERVENTIONS:
Drug: ccIIV4
  Other Names: Flucelvax
  Arms: cc IIV4
Drug: IIV4
  Other Names: Fluarix
  Arms: IIV4

SUMMARY:
This study is designed to note whether a larger safety study using quadrivalent live attenuated influenza vaccine (LAIV4) versus quadrivalent inactivated influenza vaccine (IIV4)(FLUARIX®), would be feasible in children with persistent asthma. Half of the patients in this study will receive the FLUARIX® influenza vaccine, while the other half will receive a cell cultured quadrivalent inactivated influenza vaccine (ccIIV4)(Flucelvax®) being used as a surrogate for LAIV4.

DETAILED DESCRIPTION:
The association of an increased risk in wheezing following receipt of a live-attenuated influenza vaccine in children at least 2 years of age with a prior history of asthma or wheeze remains unclear.

The Centers for Disease Control (CDC) and Prevention's Clinical Immunization Safety Assessment (CISA) planned to address a data safety gap regarding use of LAIV4 vaccine in children with asthma by conducting a 3-site randomized, non-inferiority prospective study. The main goal was to compare the safety of LAIV4 versus IIV4 in children 5-11 years with persistent asthma during the 2016-2017 influenza season. CDC and the CISA study sites developed a protocol and associated materials, and were poised to begin enrollment early during the 2016-2017 influenza season. However, after the June 22, 2016 Advisory Committee on Immunization Practices (ACIP) vote recommending against use of LAIV4 during the 2016-2017 influenza season, CDC and study investigators decided to defer implementing a study using LAIV4 during the 2016-2017 influenza season. Investigators will reconsider initiating this study during the 2017-2018 influenza season if ACIP votes to reinstate LAIV4 use or new data become available; ACIP makes recommendations annually.

The planned LAIV4 study had unique features in its design that previously had not been implemented in vaccine safety studies, including: 1) enrolling a substantial proportion of children with moderate-severe asthma 2) using digital peak flow meters and 3) collecting clinical data through multiple, complementary, measures for 42 days after vaccination. To capitalize on progress made during development of the study protocol and associated documents and procedures, CISA is proposing to carry out a study at the three sites to assess the feasibility of recruiting, enrolling, retaining, and collecting clinical data on children 5-11 years with persistent asthma of varied levels of severity in an influenza vaccine safety study. Findings from this proposed feasibility study will facilitate improving the LAIV4 study in the future if it goes forward through the CISA Project or in another venue. In 2016-2017 season, FDA approved a new influenza vaccine for use in persons aged 4 years and older, Flucelvax® Quadrivalent (ccIIV4); ACIP incorporated this vaccine into its recommendations for the 2016-2017 influenza season. Therefore ccIIV4 will be used in place of LAIV4 for this feasibility study. There is no evidence that Flucelvax® increases the risk of wheezing in asthmatic children. The feasibility study also offers an opportunity to gain some additional descriptive safety data for this new vaccine in asthmatic children.

ELIGIBILITY:
Inclusion Criteria:

* Children between 5-11 years of age, inclusive, at enrollment.
* Participant must have a current diagnosis of persistent asthma.
* Parent/legal guardian must provide written informed consent and subject must provide assent as appropriate for age prior to initiation of study procedures and according to local Institutional Review Board (IRB) requirement.
* Parent/legal guardian and subject must be willing and able to comply with planned study procedures and be available for all study visits.
* Children aged 5-8 years must have received at least 2 doses of seasonal trivalent or quadrivalent influenza vaccine prior to the current influenza season. Children 9-11 years must have received at least 1 dose of seasonal trivalent or quadrivalent influenza vaccine prior to the current influenza season.
* Is in good health, other than their asthma, as determined by medical history and targeted physical examination based on medical history.
* English or Spanish literate.
* Intention of being available for entire study period and complete all relevant study procedures, including follow-up phone calls and collection of information.

Exclusion Criteria:

* Acute illness and/or a reported oral temperature of ≥ 100.4°F within 72 hours prior to enrollment (this may result in a temporary delay of vaccination.
* Use of antipyretic medication during the preceding 24 hours that might mask a fever (temporary deferral).
* History of a severe allergic reaction (e.g., anaphylaxis) to any component of study influenza vaccines or a known allergy to eggs.
* Receipt of any licensed vaccine within 14 days (for inactivated vaccines) or 28 days (for live vaccines) prior to vaccination or planned receipt of any licensed vaccine within 42 days after vaccination.
* Receipt of current year's licensed influenza vaccine.
* Received an investigational agent (licensed or unlicensed vaccine, drug, biologic, device, blood product, or medication) in the 28 days prior to enrollment or planned receipt before 42 days after vaccination.
* Has immunosuppression as a result of an underlying illness or treatment, or use of anticancer chemotherapy or radiation therapy within the preceding 36 months.
* Has taken ≥ 20mg/day of prednisone or its equivalent, for 14 days or more within the past 28 days.
* Has know active neoplasm or a history of any hematologic malignancy.
* Has had a previous exacerbation of their asthma symptoms requiring systemic steroids within the prior 28 days, or has had a life-threatening exacerbation of asthma in the past two years (e.g. hypoxic seizure, mechanical ventilation).
* History of Guillian-Barre syndrome within 6 weeks of previous influenza vaccination.
* Has any condition that, in the opinion of the investigator, would interfere with the evaluation of the responses or would place the participant at unacceptable risk of injury.
* Has any diagnosis, current or past, of schizophrenia, bipolar disease, or other major psychiatric disorder.
* Currently taking aspirin or aspirin-containing products.

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2016-10-10 (Actual); Primary Completion 2017-02-01 (Actual); Study Completion 2017-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn M Edwards, MD, Principal Investigator — Vanderbilt Vaccine Research Program
Locations (4):
- United States (4):
  - Centers for Disease Control and Prevention, Atlanta, Georgia
  - Duke Clinical Vaccine Unit, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Vanderbilt Vaccine Research Program, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Feasibility Measures are done by the parent/guardian of the participants. Feasibility Measure data will be reported as a single group.
  Participant data (vaccine data) will be reported by the type of vaccination received.
Groups:
- ccIIV4: 0.5 mL intramuscular injection
  ccIIV4
- IIV4: 0.5 mL intramuscular injection
  IIV4
Period: Overall Study
Arm/Group | ccIIV4 | IIV4
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ccIIV4 | IIV4 | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20 | 20 | 40
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 10 | 16
  Male | 14 | 10 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 4 | 4
  Not Hispanic or Latino | 20 | 16 | 36
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 6 | 15
  White | 9 | 9 | 18
  More than one race | 2 | 5 | 7
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Feasibility Benchmark: Number of Parents That Complete the Memory Aid 1.
Description: Memory aid 1 is a diary completed by the subjects Parent. Daily symptoms, peak flow and requires the parent to record daily symptoms, peak flow, days, post-vaccination asthma clinical symptoms and symptom scores, adverse event, fever and concomitant medication administration data for 14 days (until day 15) after vaccination.
Time Frame: 15 days
Population: Feasibility Measures are done by the parent/guardian of the participants and results are not dependent on the type of vaccine received. Feasibility Measure data will be reported as a single group.
Measure: Count of Participants; unit: Participants
Groups:
- All Parents: Parents of participants from both arms
Arm/Group | All Parents
Number analyzed (Participants) | 40
Participants | 35

2. Primary Outcome: Feasibility Benchmark: Number of Parent Completing Collection of Adverse Event Data
Description: Parent will collect the following data: need for new prescription or nonprescription medications for the control of asthma, an unscheduled healthcare provider visit or consultation within 42 days after vaccination, any other clinically significant event occurring at any point during the study period. Serious Adverse Events (SAEs) will also be monitored through 42 days after vaccination and will include events that result in death, were life threatening, result in subject hospitalization or prolongation of existing hospitalization, result in persistent or significant disability or incapacity. Additionally, important medical events that may not have resulted in death, were not life threatening, or did not require hospitalization might be considered SAEs when, according to appropriate medical judgment, they jeopardize the patient or subject and require medical or surgical intervention to prevent one of the outcomes listed above.
Time Frame: Day 16 to 43
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- All Participants: Participants from both arms
Arm/Group | All Participants
Number analyzed (Participants) | 40
Participants | 37

3. Primary Outcome: Feasibility Benchmark: Number of Parents That Perform and Document All Home Digital Peak Flow Measurements
Description: Number of parents that perform and document all home digital peak flow measurements at least 11 days out of the 15-day monitoring period.
Time Frame: 15 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 40
Participants | 37

4. Primary Outcome: Feasibility Benchmark: Number of Parents That Perform and Document the Digital Peak Flow for Day 42
Description: Parent will perform and document the digital peak flow for Day 42
Time Frame: Day 42
Population: Feasibility Measures are done by the parent/guardian of the participants and results are not dependent on the type of vaccine received.. Feasibility Measure data will be reported as a single group.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 40
Participants | 37

5. Primary Outcome: Feasibility Benchmark: Number of Parents That Document Nighttime Awakenings
Description: Number of parents that document nighttime awakenings for at least 11 of the 15-day monitoring period.
Time Frame: 15 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 40
Participants | 37

6. Primary Outcome: Feasibility Benchmark: Number of Parents That Respond to Day 4 Call and Provide Requested Data
Description: Number of parents that respond to Day 4 ( -1 day or + 2 days) call and provide requested data
Time Frame: Day 3 to 6
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 40
Participants | 39

7. Primary Outcome: Feasibility Benchmark: Number of Parents That Respond to Day 8 Call and Provide Requested Data.
Description: Number of parents that respond to Day 8 (plus 2 days) call and provide requested data.
Time Frame: Day 8-10
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 40
Participants | 39

8. Primary Outcome: Feasibility Benchmark: Number of Parents That Respond to Day 15 Call and Provide Requested Data
Description: Number of parents that respond to Day 15 (minus 1 or plus 2 days) call and provide requested data
Time Frame: Day 14 to 17
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 40
Participants | 39

9. Primary Outcome: Feasibility Benchmark: Number of Parents That Respond to Day 29 Call and Provide Requested Data.
Description: Number of Parents that respond to Day 29 ( Plus 2 Days) call and provide requested data.
Time Frame: Day 29-31
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 40
Participants | 37

10. Primary Outcome: Feasibility Benchmark: Number of Parents That Respond to Day 44 Call
Description: Number of parents that respond to Day 44 ( Plus 3 Days) call and provide requested data.
Time Frame: Day 44-47
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 40
Participants | 36

11. Primary Outcome: Feasibility Benchmark: Number of Parents Completing a Satisfaction Survey
Description: Parent of each participant will be asked to complete a at the end of the study
Time Frame: 42 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 40
Participants | 36

12. Secondary Outcome: Severe Local Reactogenicity Events During the 14 Days Post-vaccination
Description: Number of severe local reactogenicity events for 14 days after vaccination between recipients of ccIIV4 and IIV4.
Time Frame: 14 days
Measure: Number; unit: number of events
Arm/Group | ccIIV4 | IIV4
Number analyzed (Participants) | 20 | 20
number of events | 0 | 2

13. Secondary Outcome: Severe Systemic Reactogenicity Events During the 14 Days Post-vaccination
Description: Number of solicited severe (not serious) systemic reactogenicity events for 14 days after vaccination between recipients of ccIIV4 and IIV4.
Time Frame: 14 days
Measure: Number; unit: number of events
Arm/Group | ccIIV4 | IIV4
Number analyzed (Participants) | 20 | 20
number of events | 1 | 1

14. Secondary Outcome: Unsolicited and Severe Adverse Events
Description: The nature and frequency of the unsolicited and Severe adverse events will be described in children receiving ccIIV4 and IIV4 during the 42 days after vaccination.
Time Frame: 42 days
Measure: Number; unit: number of events
Arm/Group | ccIIV4 | IIV4
Number analyzed (Participants) | 20 | 20
number of events
  wheezing | 1 | 0
  hand foot and mouth virus | 1 | 0

15. Secondary Outcome: Number of Asthma Exacerbations Requiring Steroids
Description: For the purpose of this study, asthma exacerbation will be defined as: any acute episode of progressively worsening shortness of breath/dyspnea, cough, wheezing, chest tightness, and/or respiratory distress during the 42 days post-vaccination (until day 43) for which the patient receives a new prescription for systemic corticosteroids..
Time Frame: 42 days
Measure: Number; unit: number of events
Arm/Group | ccIIV4 | IIV4
Number analyzed (Participants) | 20 | 20
number of events | 3 | 1

16. Secondary Outcome: Number Participants With Asthma Exacerbations Requiring Medical Attention
Description: For the purpose of this study, asthma exacerbation will be defined as: any acute episode of progressively worsening shortness of breath/dyspnea, cough, wheezing, chest tightness, and/or respiratory distress during the 42 days post-vaccination (until day 43) for which the patient seeks unscheduled medical attention (e.g., healthcare provider office or Emergency Department visit or hospitalization)
Time Frame: 42 days
Measure: Count of Participants; unit: Participants
Arm/Group | ccIIV4 | IIV4
Number analyzed (Participants) | 20 | 20
Participants | 6 | 4

ADVERSE EVENTS:
Time Frame: 42 days from vaccination
Arm/Group | ccIIV4 | IIV4
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 1/20 | 0/20
Other Adverse Events (participants affected / at risk) | 19/20 | 19/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ccIIV4 (N=20) | IIV4 (N=20)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hand foot and mouth disease (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ccIIV4 (N=20) | IIV4 (N=20)
Asthma Exacerbations (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 4 (4)
Local Reaction to Vaccine (Immune system disorders) | 19 (19) | 19 (19) — includes mild, moderate and severe local reactions
Feverish (Immune system disorders) | 4 (4) | 5 (5)
Headache (General disorders) | 7 (7) | 7 (7)
Muscles Aches (General disorders) | 2 (2) | 5 (5)
Bone Pain (General disorders) | 2 (2) | 4 (4)
Fatigue (General disorders) | 6 (6) | 12 (12)
Decrease Appetite (General disorders) | 4 (4) | 8 (8)
Stomache Ache (Gastrointestinal disorders) | 6 (6) | 7 (7)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3)
Irritability (General disorders) | 7 (7) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-19): https://cdn.clinicaltrials.gov/large-docs/93/NCT02967393/Prot_SAP_000.pdf